CLINICAL TRIAL: NCT07369700
Title: Evaluation of an mHealth-CHW Tool for Post-c-section Follow-up in Rural Rwanda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Partners in Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 25-2585; R33HD103052 (NIH); IRB25-2528 (Other: University of North Carolina Chapel Hill)
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Surgical Site Infection Following Cesarean Delivery; Cesarean Section Complications

STUDY DESIGN:
Masking Description: Random assignment - participants will be randomly assigned to an arm, and both participants and study team members will not know what the assignment is until the day the participant is to be discharged from the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care (No Intervention): Individuals randomized to this arm will receive the standard of care for women recovering from c-section in Rwanda, which is guidance to return to their nearest health center every few days for check up until advised otherwise.
- Intervention, mHealth-CHW tool (Experimental): Individuals in this arm will receive the intervention, whereby they will be followed up at postoperative days 5 and 10 at their homes by a study community health worker (sCHW) using the mHealth-CHW tool. When using this tool, individuals will be asked a series of yes-no questions inquiring about symptoms which may indicate potential post c-section complications, and have a picture of their c-section wounds captured using the tool, which would predict whether the wound is infected or not. The sCHW would then relay the guidance produced by the app, which may be that the individual can continue to recover safely at home or that they should seek help at their nearest health facility for the identified symptoms.
  Interventions: Behavioral: mHealth Community Health Worker Intervention for post-cesarean follow up

INTERVENTIONS:
Behavioral: mHealth Community Health Worker Intervention for post-cesarean follow up — Individuals will be followed up at postoperative days 5 and 10 at their homes by a study community health worker (sCHW) using the mHealth-CHW tool. When using this tool, individuals will be asked a series of yes-no questions inquiring about symptoms which may indicate potential post c-section complications, and have a picture of their c-section wounds captured using the tool, which would predict whether the wound is infected or not. The sCHW would then relay the guidance produced by the app, which may be that the individual can continue to recover safely at home or that they should seek help at their nearest health facility for the identified symptoms.
  Arms: Intervention, mHealth-CHW tool

SUMMARY:
Cesarean sections (c-sections) are one of the most common surgical procedures done globally. However, there has been an increase in the number of c-section related complications. Women who deliver via c-section are nearly twice as likely to experience a complication (not including hemorrhage) as compared to women who deliver vaginally. One of the most commonly reported postoperative complications is surgical site infections (SSIs) - in this case, an infection of the c-section wound - with the highest rates of infection globally being in African regions (11.91%). In Rwanda, patients receive verbal instructions after surgery to return to the hospital should they experience an SSI or other complication. However, there is often patient delay in identification of complications and return to care, which increases rates of morbidity (illness) and mortality (death) from post c-section complications. The investigators think that if patient follow-up after operation is improved, this may reduce the impact of complications on patient health and well-being. This research is being done to evaluate the mHealth-CHW tool developed to support comprehensive home-based follow-up by community health workers (CHWs).

Patients who have had c-section at Kirehe District Hospital will be recruited for this study, and will be randomly assigned to one of two groups: the intervention for home follow-up using the mHealth-CHW tool (referred to as Arm 1) or the standard of care (referred to as Arm 2). Individuals assigned to Arm 1 will be visited at home twice by a study CHW (sCHW) using the mHealth-CHW tool. They may be instructed to return to the health center for care based on the visit using the mHealth-CHW tool. Individuals in Arm 2 will follow the current standard of care and will be instructed to return to a health center every few days for follow-up until instructed otherwise. Regardless of the arm assignment, all participants will be instructed to return to Kirehe District Hospital 30 days after the date of their operation for a study clinic. At this study clinic they will undergo physical exam by a general practitioner (the healthcare provider who typically sees patients post c-section at the hospital level in Rwanda) and the study team will ask questions regarding financial expenditure for us to understand the rate of financial catastrophe experienced by both groups.

DETAILED DESCRIPTION:
Procedures at enrollment:

After c-section delivery and during hospitalization, eligible participants will undergo a full consent process whereby study staff will inform them of study objectives and invite the individuals to participate in the study. For this study, the investigators will prospectively enroll individuals who have delivered via c-section at Kirehe District Hospital (KDH) and are residents of Kirehe District over a nine-month window. Around the time of enrollment study staff will record demographic and routine clinical data from the patient self report and patient's charts. Participants will be randomly assigned to the intervention arm (Arm 1) or standard of care arm (Arm 2). This assignment will be contained in a numbered study packet, which additionally contains details on arm-specific follow-up, such as the follow-up plan for home visits (Arm 1) or standard of care procedures (Arm 2); general discharge instructions, including identifying signs of surgical site infection; how to contact study staff; and how to return to a health center for care or referral to KDH if a complication is suspected by a study Community Health Worker (sCHW).

Procedures at time of discharge and prior to postoperative day 30 At the time of discharge participants will receive their study packet, and their arm assignment will be revealed. Study staff will also capture wound images prior to discharge. The images are collected to help improve the technology used to predict whether a c-section wound is infected or not based on wound images.

Procedures for participants randomized to Arm 1: sCHWs will follow-up with the participants randomized to Arm 1 five days post operation (±1 day) and 10 days post operation (±1 day). sCHWs will use the mHealth-CHW tool to conduct the follow-up. During follow up, the sCHW will be guided by the mHealth-CHW tool to ask a series of yes-no questions identifying whether the participant is experiencing symptoms which may be related to post c-section complications, then they will be prompted to take a picture of the participant's c-section wound, which the app will use to predict whether the wound is infected or not. If any potential complications are detected by the mHealth-CHW tool the sCHW will advise the participant to seek care at their nearest health center or the hospital. sCHWs will use a paper form to track implementation measures related to process and phone functionality. To measure time-to-diagnosis for the mHealth-CHW tool the complication must be confirmed and documented at a health center.

Procedures for participants randomized to Arm 2: Participants randomized to Arm 2 will follow the current standard of care for post-c-section follow-up. In the current standards of care following c-section in Rwanda, women who have had c-section are advised to return to a health center every 3-5 days after discharge until instructed otherwise by health center staff.

For both arms, any complications identified at the health centers will be logged by nurses in study registers. Nurses at these health centers will log any complication identified among c-section patients during the nine-month study window, with details on the complication, date, and treatment/referral plans.

Follow-up:

All participants will be asked to return to the hospital 30 days after their operation (±7 days) for a special study clinic held on Wednesdays; participants will receive a voucher to cover transport costs to the hospital and will be compensated for their time in accordance with the Rwanda National Ethics Committee (RNEC) guidelines. The visit will be conducted by a Kirehe-based general practitioner (the healthcare provider who typically sees patients post c-section at the hospital level in Rwanda) who will perform a full clinical and physical exam. A study data collector will document any post-c-section complications detected by the general practitioner. A study nurse will then interview participants to record post-discharge activities, including health seeking behaviors and any diagnoses or care instructions received outside of the home and study clinic visits. The study nurse will review health center registers to confirm participant reports of these visits or to identify any visits that were not reported by participant, and capture a wound image. All women will report health care expenditures using a financial survey questionnaire adapted from the Program for Global Surgery and Social Change National Surgical Obstetric Anesthesia Plan surgical indicator questionnaire. This will be used for us to understand the rate of financial catastrophe (spending more than 10% of the family's annual household expenditures on post c-section follow-up) experienced by both groups.

There are two study clinics that fall within the study clinic window (30 days post-operation, ±7 days). The participant will be scheduled for the first. If they miss this visit, they will be rescheduled for the second visit. If the participant misses the two visits, they will be considered lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Had cesarean delivery at Kirehe District Hospital (KDH), Rwanda; resident of Kirehe District, Rwanda

Exclusion Criteria:

* Did not have cesarean delivery at KDH; not resident of Kirehe District; residence in Mahama refugee camp

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Time-to-diagnosis for complications | From enrollment to the time of participation at the study clinic (30 days post operation)
  For time-to-diagnosis, for each woman with an identified complication, time-to-diagnosis will be date from cesarean to date of diagnosis, either at the health center or at the hospital study clinic visit. Complications after the study clinic visit will be excluded. Assessments at the health center and/or study clinic will provide a clinical validation of the findings.
Completion of intervention steps (follow-up using mHealth-CHW tool) | 5 (±1 day) and 10 (±1 day) days post c-section
  For completion of intervention steps in mHealth-CHW tool, the investigators will report the proportion of visits with all steps completed. A visit is considered complete if all steps above were successfully completed within one hour of the study community health worker (sCHW) arriving at the home. The steps included are:
  Being able to find patients home. Participant willing to have physical exam by sCHW. The sCHW completed the basic assessment as guided by the tool. The sCHW completed the photo-based SSI diagnosis as guided by the tool. The sCHW provided general counseling and follow-up instructions as guided by the tool.
  The full home screening was completed. Phone could turn on. Phone did not shut down during interaction. Phone maintained charge. If needed, was the phone successfully recharged in field. Data from screening successfully stored.

SECONDARY OUTCOMES:
Cesarean-associated complications (mHealth-CHW tool) | From enrollment to the time of participation at the study clinic (30 days post operation)
  Secondary outcomes will include presence of cesarean-associated complication, and complication identification by the mHealth-CHW tool screening. Evaluation of surgical site infection will be conducted using a machine learning (ML) algorithm within the mHealth-CHW tool, and symptom mapping will be used to link symptoms with specific post-cesarean conditions.
Financial catastrophe | From enrollment to the time of participation at the study clinic (30 days post operation)
  The investigators will document whether or not the c-section was financially catastrophic, defined as spending more than 10% of the family's annual household expenditures on follow-up. At the study clinic all women will report health care expenditures and general financial resources using a financial survey questionnaire adapted from the Program in Global Surgery and Social Change National Obstetric Anesthesia Plan surgical indicator questionnaire, which has been previously used in this setting (Niyigena et al. 2022). The finding will be reported as the proportion of women who experienced financial catastrophe.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Hedt-Gauthier, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kirehe District Hospital, Kirehe, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared in a public repository, if approved by the Rwanda government.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months after and continuing for 36 months following publication
Access Criteria: If approved by Rwanda government, data will be made available in a publicly available repository.